CLINICAL TRIAL: NCT04542109
Title: READyR: A Remote Assessment and Dynamic Response Intervention to Support Couples in Planning for Changing Dementia Care Needs
Brief Title: REmote Assessment and Dynamic Response Intervention
Acronym: READyR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lyndsey Miller, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional 16-2; P30AG024978-16 (NIH)
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Dementia; Alzheimer Disease; Relationship, Marital; Caregiver Stress Syndrome
Keywords: Needs Assessment; Family Caregiver; Technology; Remote Monitoring; Care Values; Aging-in-place
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Dyads will be randomized (assigned by chance) to one of two groups: 1) READyR A or 2) READyR B (Wait List Control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- READyR A (Experimental): Group A will start the READyR intervention immediately after the baseline Session 1. The READyR program consists of a 3-session, values-based needs assessment intervention designed to match objectively-assessed in-home activity patterns with subjective reports of participants' care values. The goal of the intervention is to address unmet dementia-related care needs and help couples prepare for the future, and reduce strain on their relationship, and help maintain their health and well-being. Session 2 will occur approximately 3 weeks after Session 1, and Session 3 will occur approximately 3 weeks after Session 2. Session 3 also includes follow-up assessments.
  Interventions: Behavioral: READyR A
- READyR B (wait list comparison) (Active Comparator): Group B - the wait list comparison group - will have a 60-minute support session (comparator intervention) about 3 weeks after the baseline Session 1. The support session will include general information about dementia-related care needs that does not take into account the individual participant's care values or objective in-home activity patterns. They will also receive a check-in call approximately 3 weeks later, with follow-up assessments. Group B will begin the READyR intervention sessions following completion of follow-up assessments.
  Interventions: Behavioral: READyR B

INTERVENTIONS:
Behavioral: READyR A — Two active sessions to conduct an individually-tailored dementia-related needs assessment, incorporating the participant's care values and objective data from remote in-home monitoring.
  Other Names: SHARE-sense
  Arms: READyR A
Behavioral: READyR B — Active comparator. Two sessions to deliver general information about dementia-related care needs.
  Arms: READyR B (wait list comparison)

SUMMARY:
The purpose of the READyR study (originally called SHARE-sense) is to redevelop and test an intervention program to remotely assess for changing dementia-related care needs.

DETAILED DESCRIPTION:
Unmet dementia-related care needs are highly prevalent, and are detrimental to the care dyad's (person with dementia and their family care partner) health, safety, mortality, and likelihood of nursing home placement. The first phase of this study involves redevelopment of the intervention program into a 3-session values-based needs assessment intervention (delivered over 6 weeks) designed for early-stage persons with dementia and their primary family caregiver (i.e. spouse or partner). A secondary data analysis and focus groups will be conducted in order to complete the redevelopment phase. Objective digital data on behavioral patterns (from sensors and wearables) will be incorporated into a needs assessment that will allow for dynamic tailoring of the READyR program to new and unforeseen care needs.

People who voluntarily decide to participate in this study will be asked to participate in three sessions: Session 1 for baseline assessments gathered from all participants (including remote in-home monitoring), Session 2 for discussing the participant's care values and their alignment with current patterns of activities (assessed by remote monitoring) in the home, and Session 3 for addressing current dementia related care needs and setting goals for the future.

Participants who complete this study will be offered participation in a follow-up monitoring period to further study the possibilities for dynamic tailoring of their dementia-related needs assessment.

ELIGIBILITY:
Persons with Dementia

Inclusion:

1. 62 years or older;
2. Able to identify a family care partner over age 20 who is living with you and will also consent to fully participate in the study;
3. Probable or confirmed diagnosis of mild cognitive impairment or early-stage dementia
4. Age and education adjusted MOCA score > 15 (at most recent measurement by parent study) corresponding to early to moderate stage dementia

Exclusion:

1. Inability to speak English or read printed materials in English
2. Conditions that would limit participation at entry to study (e.g. visual or hearing impairments prohibiting reading and discussing the intervention materials);
3. Any uncontrolled medical condition that is expected to preclude completion of the study, such as late stage cancers.

Family Care Partners

Inclusion:

1. 21 years or older;
2. Self-identifying as a family member and care partner residing with the PwD participant;

Exclusion:

1. Inability to speak English or read printed materials in English
2. Conditions that would limit participation at entry to study (e.g. visual or hearing impairments prohibiting reading and discussing the intervention materials);
3. Any uncontrolled medical condition that is expected to preclude completion of the study, such as late stage cancers.

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Mean difference effect sizes for pre-post change the care dyad's preparation for future care needs | Baseline, 6 weeks, 12 weeks
  The Preparation for Future Care Needs Scale (Short Form) assesses the degree to which an individual has engaged in planning for future care needs in late life using 15 items and 5 subscales representing distinct planning processes (awareness, gathering information, decision making, concrete planning, avoidance). Items are scored on a 5 point Likert scale with higher scores indicating greater preparation for future care needs. Sorensen, S., Chapman, B. P., Duberstein, P. R., Pinquart, M., & Lyness, J. M. (2017). Assessing future care preparation in late life: Two short measures. Psychol Assess, 29(12), 1480-1495.
Mean difference effect sizes for pre-post change in the care dyad's relationship quality | Baseline, 6 weeks, 12 weeks
  The Dyadic Relationship Scale assesses the positive dyadic interactions and negative dyadic strain experienced by caregivers (11 items) and care recipients (10 items). Items are averaged for a summary score that ranges from 0 to 3, with higher scores indicating more positive interactions in the relationship, or more relationship strain, respectively. Sebern, M.D. & Whitlatch, C.J. (2007). Dyadic Relationship Scale: A measure of the impact of the provision and receipt of family care. The Gerontologist, 47(6), 741-751.

SECONDARY OUTCOMES:
Mean difference effect sizes for pre-post change in care-related strain | Baseline and weekly for 12 weeks
  Subjective strain from caregiving will be assessed among family care partners at baseline and follow-up assessments using the Zarit Burden Interview (ZBI), short-form (12 items). Scores range from 0-48 with higher scores indicating a greater degree of strain from providing care.
Mean difference effect sizes for pre-post change in quality of life | Baseline, 6 weeks, and 12 weeks
  The Quality of Life: Alzheimer's Disease Scale assesses individual perceptions of quality of life (from poor to excellent) across 13 items. Items are averaged for a summary score of 1 to 4, higher scores indicating greater degree of quality of life. Logsdon, R. G., Gibbons, L. E., McCurry, S. M., & Teri, L. (1999). Quality of Life in Alzheimer's Disease: Patient and Caregiver Reports. Journal of Mental Health and Aging, 5(1), 21-32.
Mean difference effect sizes for pre-post change in concealment of emotions. | Baseline, 6 weeks, and 12 weeks
  The Emotional Intimacy Disruptive Behavior Scale (8 items) assesses the frequency of engagement in behaviors to conceal emotions about an illness from one's partner. Druley, J. A., Stephens, M. A. P., & Coyne, J. C. (1997). Emotional and physical intimacy in coping with Lupus: Women's dilemmas of disclosure and approach. . Health Psychology, 16, 506-514.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsey M Miller, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available upon request to our Alzheimer's Disease Research Center
Time Frame: Data will become available after completion of study and after publication of primary study aims.
Access Criteria: Requests need to made to the PI at the Oregon Alzheimer's Disease Research Center (OARDC). A short data request form will need to be submitted to the OADRC

REFERENCES:
- [Derived] Miller LM, Solomon DN, Whitlatch CJ, Hiatt SO, Wu CY, Reynolds C, Au-Yeung WM, Kaye J, Steele JS. The Remote Assessment and Dynamic Response Program: Development of an In-Home Dementia-Related Care Needs Assessment to Improve Well-Being. Innov Aging. 2022 Feb 7;6(2):igac006. doi: 10.1093/geroni/igac006. eCollection 2022. PMID 35402736